CLINICAL TRIAL: NCT00016107
Title: A Phase II Study Of Estramustine, Docetaxel, And Bevacizumab (IND # 7921, NSC # 704865) In Men With Hormone Refractory Prostate Cancer
Brief Title: Combination Chemotherapy Plus Bevacizumab in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-02962; CALGB-90006; CDR0000068595; U10CA031946 (NIH)
Record Dates: First submitted 2001-05-06; First posted 2003-06-10 (Estimated); Last update posted 2013-06-05 (Estimated); Status verified 2013-06

CONDITIONS: Adenocarcinoma of the Prostate; Hormone-resistant Prostate Cancer; Recurrent Prostate Cancer; Stage IV Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Estramustine; Docetaxel; Bevacizumab

ARMS (1):
- Treatment (chemotherapy, bevacizumab) (Experimental): Patients receive oral estramustine 3 times daily on days 1-5 and docetaxel IV over 1 hour followed by bevacizumab IV over 30-90 minutes on day 2. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: estramustine phosphate sodium; Drug: docetaxel; Biological: bevacizumab; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: estramustine phosphate sodium — Given orally
  Other Names: EM; Emcyt; Estracyt; Ro 22-2296/000
Drug: docetaxel — Given IV
  Other Names: RP 56976; Taxotere; TXT
Biological: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Phase II trial to study the effectiveness of combination chemotherapy plus monoclonal antibody therapy in treating patients who have metastatic prostate cancer that has not responded to previous hormone therapy. Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Monoclonal antibodies such as bevacizumab may stop the growth of cancer cells by stopping blood flow to the tumor. Combining monoclonal antibody therapy with chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine time to objective progression, response rate (objective and PSA response) and duration of response in men with hormone refractory prostate cancer treated with estramustine, docetaxel and bevacizumab.

II. To determine the toxicity of this regimen in men with hormone refractory prostate cancer.

III. To study the relationship of baseline VEGF levels in urine and plasma and changes in these levels to response and duration of response to treatment with bevacizumab, docetaxel and estramustine.

OUTLINE:

Patients receive oral estramustine 3 times daily on days 1-5 and docetaxel IV over 1 hour followed by bevacizumab IV over 30-90 minutes on day 2. Treatment repeats every 21 days in the absence of disease progression or unacceptable toxicity.

Patients are followed at least every 3 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically documented adenocarcinoma of the prostate with progressive systemic (metastatic) disease despite castrate levels of testosterone due to orchiectomy or LHRH agonist (which must be continued); castrate levels of testosterone must be maintained
* At the time of enrollment, patients must have evidence of metastatic disease, either:

  * Measurable disease (with any PSA) OR
  * Non-measurable disease with PSA >= 5 ng/ml; patients with PSA >= 5 ng/ml only are not eligible DEFINITION OF MEASURABLE DISEASE/TARGET LESIONS
  * Any lesion that can be accurately measured in at least one dimension (longest diameter to be recorded) as >= 20 mm with conventional techniques: 1) physical exam for clinically palpable lymph nodes and superficial skin lesions, 2) chest X-ray for clearly defined lung lesions surrounded by aerated lung OR those lesions measured as >= 10 mm with a spiral CT scan or MRI
  * Measurable lesions (up to a maximum of 10 in number) representative of all organs involved to be identified as target lesions; the sum of the longest diameters (LD) for all target lesions will be calculated and reported as baseline sum LD

    * If measurable disease is confined to a solitary lesion then its neoplastic nature will need to be confirmed by histology
    * Ultrasound may not be used to measure tumor lesions that are not easily accessible clinically DEFINITION OF NON-MEASURABLE DISEASE/NON-TARGET LESIONS
  * Non-target lesions include all other lesions, including small lesions with longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan and truly non-measurable lesions, which include:

    * Bone lesions
    * Pleural or pericardial effusions, ascites
    * CNS lesions, leptomeningeal disease
    * Irradiated lesions, unless progression documented after RT
* Patients must have demonstrated evidence of progressive disease since the most recent change in therapy; progressive disease is defined as any one of the following (measurable disease, bone scan, or PSA progression):

  * MEASURABLE DISEASE PROGRESSION: Objective evidence of increase > 20% in the sum of the longest diameters (LD) of target lesions from the time of maximal regression or the appearance of one or more new lesions
  * BONE SCAN PROGRESSION: Appearance of one or more new lesions on bone scan attributable to prostate cancer along with a PSA >= 5 ng/ml will constitute progression
  * PSA PROGRESSION: An elevated PSA (at least >= 5 ng/ml) which has risen serially from baseline on two occasions each at least one week apart. If the confirmatory PSA (#3) value is less (i.e., #3b) than screening PSA (#2) value, then an additional test for rising PSA (#4) will be required to document progression
* Failure despite standard androgen deprivation therapy
* Flutamide and megestrol acetate (any dose) must be discontinued at least 4 weeks prior to registration; bicalutamide and nilutamide must be discontinued at least 6 weeks prior to registration. If improvement following antiandrogen withdrawal is noted, progression must be established using the criteria above; primary testicular androgen suppression (e.g., with an LHRH analogue) should not be discontinued
* At least 4 weeks since any hormonal therapy, including ketoconazole, aminoglutethimide, systemic steroids (any dose), megestrol acetate (any dose)
* No prior cytotoxic chemotherapy, including estramustine or suramin
* No prior anti-angiogenesis agents, including thalidomide and bevacizumab
* >= 4 weeks since major surgery and fully recovered
* >= 4 weeks since any prior radiation and fully recovered
* >= 8 weeks since the last dose of strontium-89 or Samarium
* Patients receiving bisphosphonate therapy prior to initiating protocol treatment must have received bisphosphonates for at least 1 month and have progressive disease despite this therapy
* CTC (ECOG) performance status: 0-2
* No myocardial infarction or significant change in anginal pattern within one year or current congestive heart failure (NYHA Class 2 or higher)
* No deep venous thrombosis or pulmonary embolus within one year. No need for full-dose oral or parenteral anticoagulation; daily prophylactic aspirin is allowed
* No clinically significant peripheral neuropathy
* Granulocytes >= 1500/ul
* Platelet count >= 100,000/ul
* Creatinine =< 1.5 x upper limit of normal
* Bilirubin =< 1.0 x upper limit of normal
* AST =< 1.5 x upper limits of normal
* Urinalysis =< 1 + protein on dipstick
* PSA >= 5 ng/ml (if non-measurable disease)
* Serum Testosterone =< 50 ng/ml for patients who have not had bilateral orchiectomy

Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2001-06; Primary Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Time to objective progression | From the initiation of treatment to the date of progressive disease, assessed up to 2 years
  The Kaplan-Meier method will be used to estimate the time to disease progression.
Response rates (PSA and objective) | Up to 2 years
  Response rates will be analyzed using both objective (CR and PR) and serological parameters. The Kaplan-Meier method will be used to estimate the response (objective and PSA) duration.
Toxicity as assessed by the National Cancer Institute Common Terminology Criteria for Adverse Events version 2.0 | Up to 2 years

SECONDARY OUTCOMES:
Overall survival | Up to 2 years
  The Kaplan-Meier method will be used to estimate the overall survival.
Duration of response | From the date of the first CR or PR to the date that the patient had progressive disease, assessed up to 2 years
  Duration of PSA response is the date from the first 50% decline (or 75% decline) in PSA to the date when the patient met the criteria for progressive disease.

CONTACTS AND LOCATIONS:
Overall Officials: Joel Picus, Principal Investigator — Cancer and Leukemia Group B
Locations (1):
- Cancer and Leukemia Group B, Chicago, Illinois, United States